CLINICAL TRIAL: NCT01956851
Title: Hospital Based Pilot Study: Association of Kisspeptin Levels With Insulin Secretion in Diabetes Mellitus
Brief Title: Association of Kisspeptin Levels With Insulin Secretion in Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Ganga Care Hospital, Nagpur (Other)
Responsible Party: Principal Investigator, DR MAMTA JOSHI, CONSULTANT PHYSICIAN, Ganga Care Hospital, Nagpur
Other Study IDs: CARE/REF/IR/KPT/03/13
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus
Keywords: insulin, kisspeptin, GLP 1
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal Healthy: Normal Healthy: includes healthy patients eligible for enrolment,
- Diabetics on Oral Hypoglycemic Agents: Diabetics on Oral Hypoglycemic Agents: includes diabetic patients on oral diabetic drug therapy with all eligibility criterion fulfilled,
- Diabetics on Insulin Therapy: Diabetics on Insulin Therapy: includes diabetic patients on insulin therapy with all eligibility criterion fulfilled

SUMMARY:
Since the discovery of kisspeptin as a "gate-keeper" of hypothalamo-pituitary-gonadal axis, there has been tremendous interest in the molecule. The relevance of kisspeptin as regulatory molecule for the reproductive system has been well documented in significant number of trials. (1, 2) This leads to the possibility that kisspeptin could be involved in an equally pivotal role in the other sites, where it is located, namely pancreas.

While various animal experiments have suggested that kisspeptins regulate insulin secretion, we do not know if this is also true in humans. The investigators hypothesize that kisspeptin levels are significantly low in individuals who have low endogenous insulin secretion.

While various animal experiments have suggested that kisspeptins regulate insulin secretion, the investigators do not know if this is also true in humans. Investigators hypothesize that kisspeptin levels are significantly low in individuals who have low endogenous insulin secretion.

Thus investigators are conducting this study to understand the link between endogenous insulin secretion and kisspeptin levels among individuals with various levels of insulin secretory defect as seen in diabetics. Investigators believe that this will help understand the physiologic mechanisms, and kisspeptin based insulin regulation among individuals with diabetes mellitus.

DETAILED DESCRIPTION:
INTRODUCTION:

Since the discovery of kisspeptin as a "gate-keeper" of hypothalamo-pituitary-gonadal axis, there has been tremendous interest in the molecule. Kisspeptins are a group of peptides derived from the kiss gene, which share a common C-terminal decapeptide with an arginine-phenylalanine residue at the amino terminal.(1, 2) These peptides and their target receptor GPR54 are highly expressed in hypothalamus, anterior pituitary, islets of langerhans, and gonads. (2-5) The relevance of kisspeptin as regulatory molecule for the reproductive system has been well documented in significant number of trials. (6, 7) This leads to the possibility that kisspeptin could be involved in an equally pivotal role in the other sites, where it is located, namely pancreas.

Investigators have demonstrated that kisspeptin plays a role in regulating beta cell activity.(8) Despite previous conflicting results suggesting glucose mediated insulin secretion and insulin inhibition in different studies,(9, 10) current evidence favours role of kisspeptin in glucose mediated insulin secretion.(11) One of earliest evidence of relation of insulin resistance with falling kisspeptin levels was demonstrated by Panidis et al in 2006.

While various animal experiments have suggested that kisspeptins regulate insulin secretion, we do not know if this is also true in humans. The investigators hypothesize that kisspeptin levels are significantly low in individuals who have low endogenous insulin secretion.

Thus investigators plan this study to understand the link between endogenous insulin secretion and kisspeptin levels among individuals with various levels of insulin secretory defect as seen in diabetics. We believe that this will help understand the physiologic mechanisms, and kisspeptin based insulin regulation among individuals with diabetes mellitus.

Researchers have also noted that the mechanism of stimulating glucose induced insulin release, is similar to the GLP1(Glucagon like peptide) action.(10) It would be interesting to ascertain a correlation between the two peptides with potentially similar action in insulin physiology. Leptin has been shown to alter kiss-1 expression in animal models. Establishing a link between leptin levels with kisspeptin in humans would help us identify further potential therapeutic targets involved in the multisystem manifestations of diabetes.(12)

AIMS AND OBJECTIVES:

1: To explore the association between levels of fasting insulin and kisspeptin levels, in diabetes mellitus.

2. To explore association between Obesity and Kisspeptin levels. 3. To explore the association between kisspeptin and GLP-1 levels. 4. To explore the association of leptin and kisspeptin levels.

RESEARCH QUESTION:

In a population of adults attending the outpatient diabetes and medicine clinic of a tertiary care hospital, Do those with diabetes mellitus as compared to those without diabetes mellitus, have progressively lower kisspeptin levels, and is this gradient in Kisspeptin levels related to fasting endogenous insulin secretion. Investigators hypothesize low Kisspeptin levels to be associated with low insulin secretion.

STUDY TYPE- STUDY DESIGN: Cross-sectional study Ethical approval for the trial protocol obtained from the institute's ethics committee of Care Hospital, Nagpur, India

Subjects and Methods The study will be conducted in CARE Hospital, Nagpur from 1 September 2013- 31 November 2013. Patients will be selected to enter the study, in such a way that every patient presenting to the diabetes and medicine clinic will be screened in the study and patients fulfilling inclusion criteria will be recruited in the study.

Study population:

Total of 60 patients will be included in the study. Investigators plan to include Diabetics without exogenous insulin supplementation, Diabetics with exogenous insulin supplementation and normal healthy cohorts, 20 in each group.

Methods:

The investigators will screen all patients who are referred to them after fulfilling the inclusion and exclusion criteria in the study. Written informed consent will be obtained from all participants. The patients included in the study will be administered a standardized questionnaire to record socio-demographic characteristics, details of diabetes management, history of PCOD (Polycystic Ovarian Disease), history of hypogonadism or any obvious sexual dysfunction drug history. A general examination for BMI (Body mass index), waist hip ratio and Blood pressure would be performed. Blood samples will then be withdrawn (8 ml : 2ml fluoride tube, 2ml EDTA (ethylenediaminetetraacetic acid ), 4 ml plain tube) after overnight fasting for creatinine, fasting blood glucose, fasting insulin, C-peptide levels, HbA1C (glycosylated haemoglobin), LH (luteinizing hormone), FSH (Follicle stimulating hormone), and kisspeptin levels. In female patients samples will be collected between day 3 to day 6 of a normal menstrual cycle. After a usual meal as regularly taken by the patient, samples (8ml: 2ml fluoride, 4ml EDTA and 2 ml plain tube) for post-prandial blood glucose level, insulin level, leptin level, GLP-1 level and kisspeptin levels will be collected. The blood samples for creatinine, glucose (pre and post), insulin levels, HbA1C, LH and FSH will be analysed immediately in the laboratory. The blood samples for kisspeptin levels, GLP-1, leptin levels will be collected in a separate EDTA tube, centrifuged for 15 min at 4 degree and plasma will be stored separately in a deep freezer at -70 degree. The concentration of kisspeptin will be measured using Kiss¬peptin-10 (Metastin [45-54]-Amide) and competitive enzyme immunoassay (Kit# EK-048-56, Phoenix Pharmaceuticals, Inc., Burlingame, CA, USA). Leptin (Human) ELISA Kit Protocol (Cat. No.: EK-003-12, Phoenix Pharmaceuticals) will be used for serum leptin levels. GLP-1 (7-36)-Amide (Human,Rat, Mouse) EIA (enzymeimmunoassay) Kit (Catalog # EK-028-11, Phoenix Pharmaceuticals) will be used for testing GLP 1 levels. The method given in the product insert will be used for the assays.

Power analyses There is no similar study done to help us predict the power of study. As the investigators did not have previous estimates no formal power calculation was undertaken. The investigators randomly decided to take 60 patients in the study, 20 in each arm.

Data analysis All data will be entered using MS excel. Researchers will perform a descriptive statistical analysis of the baseline data. The analyst, who will be blinded to the laboratory results, will compare the outcome measure using Pearsons coefficient of correlation. All statistical analysis will be done using SPSS software (v.16.0 SPSS, Inc., Chicago, IL) Dissemination The results of this trial are expected to provide evidence and clinically relevant information the relation between kisspeptin and diabetes.

Risks of participation The investigators believe there is no additional risk for the participants included in the study.

Competing interests The authors declare that they have no competing interests.

ELIGIBILITY:
Inclusion criteria- Patient's between 25-45 yrs, belonging to either sex.

Exclusion criteria-

* Patients of age group more than 45 yrs and below 25 years
* Pregnant or lactating or post menopausal females.
* Females with irregular menstrual cycles or galactorrhea
* Patients on medications interfering with hormonal functions
* Patients with history suggestive of gonadal dysfunction (hypogonadism primary or secondary)
* Patients with polycystic ovarian disease (PCOD)
* Patients with chronic kidney disease with GFR (Glomerular Filtration rate) <60ml/min
* Patients receiving gonadal therapy in the form of GnRH (gonadotropin-releasing hormone) agonist or antagonist, estrogen, progesterone or testosterone preparations
* Patients not willing to give informed consent

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients entering medical and diabetes out patient clinics
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
correlation of kisspeptin levels with GLP 1 | 2 hours post meal

CONTACTS AND LOCATIONS:
Overall Officials: Mamta N Joshi, Principal Investigator — Ganga CARE Hospital
Locations (1):
- Ganga Care Hospital, Nagpur, Maharashtra, India